CLINICAL TRIAL: NCT05534646
Title: Phase II Study of Apalutamide With Carotuximab in Metastatic, Castration-Resistant Prostate Cancer
Brief Title: Study of Apalutamide With Carotuximab in Metastatic, Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Edwin Posadas, MD (Other)
Collaborators: Enviro Therapeutics, Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Edwin Posadas, MD, Co-Director, Experimental Therapeutics Program, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021-06-Posadas-APA105
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: Prostate cancer; Castration-resistant; CRPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; carotuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apalutamide monotherapy (Active Comparator): After progression, subjects will crossover to combination therapy
  Interventions: Drug: Apalutamide
- Combination therapy (Apalutamide + Carotuximab) (Experimental)
  Interventions: Drug: Apalutamide; Drug: Carotuximab

INTERVENTIONS:
Drug: Apalutamide — Standard of care Apalutamide 240 mg administered orally and daily on Days 1-28 of every 28 day cycle
Drug: Carotuximab — Carotuximab administered intravenously at the following doses:
  Cycle 1 Day 1: 3 mg/kg Cycle 1 Day 4: 7 mg/kg Cycle 1 Day 8: 10 mg/kg Cycle 1 Day 15: 10 mg/kg Cycle 1 Day 22: 10 mg/kg Cycle 2 Day 1: 15 mg/kg Cycle 2 Day 15: 15 mg/kg Cycle 3+ Day 1: 15 mg/kg After completion of cycle 2, dosing of carotuximab will continue at a q4 week schedule using the 15 mg/kg dose.
  Arms: Combination therapy (Apalutamide + Carotuximab)

SUMMARY:
This is an open-label, multi-site study of apalutamide with carotuximab in patients who have progressed on androgen receptor signaling inhibitor (ARSI) therapy. This study will begin with a safety assessment in the first 10 subjects (part 1: Safety Lead-in). If the combination is deemed safe, the trial will proceed to the Phase II stage. The purpose of this study is to compare progression free survival (PFS) between patients receiving apalutamide and apalutamide + carotuximab using Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and Prostate Cancer Working Group 3. The secondary objectives are to describe adverse events related to the intervention, overall response rate (ORR), proportion of patients resistant to apalutamide that benefit from the addition of carotuximab, and to determine the ORR, radiographic PFS, and biochemical PFS in the overall population.

ELIGIBILITY:
Inclusion Criteria:

* History of castration-resistant prostate cancer with rising PSA (prostate-specific antigen) on a contemporary ARSI (Androgen receptor (AR) signaling inhibitor: abiraterone, enzalutamide, darolutamide). Bicalutamide, nilutamide, and flutamide will not be considered as contemporary ARSIs
* Patient must have had 1 and can have up to 2 prior AR targeted therapy with the exception of apalutamide.
* Patients must decline or be ineligible for taxane therapy in the opinion of the treating physician.
* All patients must agree to use an adequate method of contraception, in the opinion of the treating investigator, while on protocol treatment and for 3 months after the last dose of protocol treatment (apalutamide and/or carotuximab)

Exclusion Criteria:

* Non-PSA producing prostate cancers such as small cell prostate cancers or those prostate cancers which exhibit radiographic progression without PSA rise
* Prior use of apalutamide
* Other prior malignancy requiring active anticancer therapy
* Prior exposure to carotuximab or any CD105 targeted antibody
* Active bleeding or pathologic medical conditions that carries a high bleeding risk
* A known diagnosis of Osler-Weber-Rendu syndrome

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (rPFS) between patients receiving apalutamide and apalutamide + carotuximab | From the start of study treatment until documented progression, or death due to any cause, up to 30 days of follow-up after end of treatment.
  From the start of study treatment until documented progression, per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and Prostate Cancer Working Group 3, or death due to any cause.

SECONDARY OUTCOMES:
Incidence of Adverse events (grade 3 or higher) related to carotuximab and apalutamide | From start of study treatment through 4 weeks on treatment
  Grade 3 or above treatment related adverse events as assessed per NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Overall radiographic response rate (ORR) of the combination of apalutamide + carotuximab | From the start of combination study treatment until documented progression, or death due to any cause, up to 30 days of follow-up after end of treatment.
  Participants of the combination of apalutamide + carotuximab, with confirmed complete response (CR) or partial response (PR) per RECIST v.1.1 and Prostate Cancer Working Group 3
Proportion of patients resistant to apalutamide benefit from the addition of carotuximab | From the start of combination therapy study treatment until documented progression, or death due to any cause, up to 30 days of follow-up after end of treatment.
  Participants of the monotherapy group that crossover to combination therapy at progression, with confirmed complete response (CR) or partial response (PR) per RECIST v.1.1 and Prostate Cancer Working Group 3
Overall radiographic response rate (ORR) in the overall population | From the start of study treatment until documented progression, or death due to any cause, up to 30 days of follow-up after end of treatment.
  Determined by confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and Prostate Cancer Working Group 3
To determine the radiographic progression free survival (rPFS) in the overall population | From the start of study treatment until documented progression, or death due to any cause, up to 30 days of follow-up after end of treatment.
  From the start of study treatment until documented progression, per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and Prostate Cancer Working Group 3, or death due to any cause.
To determine the biochemical PFS (by PCWG3) in the overall population | From the start of study treatment until documented progression, or death due to any cause, up to 30 days of follow-up after end of treatment.
  From the start of study treatment until documented progression, per Prostate Cancer Working Group 3, or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Posadas, MD FACP, Principal Investigator — Cedars-Sinai Medical Center
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Huntsman Cancer Institute and Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No